CLINICAL TRIAL: NCT03588026
Title: Investigational Product ; Coversin. Phase III Safety and Efficacy in Three-Part, Two-Arm, Randomised Open Label Evaluation in Patients With Paroxysmal Nocturnal Haemoglobinuria (PNH)
Brief Title: Treating Paroxysmal Nocturnal Haemoglobinuria Patients With rVA576
Acronym: CAPSTONE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AKARI Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK580
Record Dates: First submitted 2018-06-01; First posted 2018-07-17 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2020-11

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 - 9 months of treatment (rVA576 plus SOC) (Experimental): 6 months (SOC plus rVA576), Followed by a further 3 months of (SOC plus rVA576).
  Interventions: Drug: rVA576; Other: Standard of care (SOC)
- Arm 2 - 6 months on SOC (Experimental): 6 months on SOC only. Followed by 3 months (SOC plus rVA576).
  Interventions: Drug: rVA576; Other: Standard of care (SOC)

INTERVENTIONS:
Drug: rVA576 — 6 months of treatment, rVA576 plus SOC. Followed by a further 3 months of rVA576 plus SOC. In total, 9 months on rVA576 plus SOC.
Other: Standard of care (SOC) — 6 months on SOC followed by 3 months of treatment with rVA576 plus SOC. In total, 3 months on rVA576 plus SOC.

SUMMARY:
rVA576 for patients with Paroxysmal Nocturnal Hemoglobinuria (PNH).

DETAILED DESCRIPTION:
rVA576, a small protein complement C5 inhibitor which prevents the cleavage of C5 by C5 convertase into C5a and C5b, will be used in an open label, non-comparative clinical trial in patients with PNH.

Patients will be treated with rVA576 by daily subcutaneous injection in order to determine the safety and efficacy of the drug in these circumstances.

If satisfactory control of the PNH is achieved, and at the discretion of the Principal Investigator (PI), patients will have the option of remaining on rVA576 and being entered into the long term follow-up study.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to give informed consent to treatment with rVA576
2. Diagnosed with paroxysmal nocturnal haemoglobinuria (PNH)
3. Have not received any complement inhibitor within the 4 months prior to screening
4. ≥ 18 years of age at the time of screening
5. Weight ≥50kg
6. Complete transfusion medical history for 12 months
7. Transfusion dependent
8. LDH ≥1.5 x the ULN
9. Willing to receive appropriate prophylaxis against Neisseria meningitidis infection, by both immunisation and continuous or intermittent antibiotics
10. Willing to avoid prohibited medications such as other complement inhibitors and chemotherapeutic agents
11. Patients must agree to avoid pregnancy and fathering children from the time of signing the Informed Consent Form until 90 days after the last dose of rVA576.
12. Patients who are on erythropoietin and/or immunosuppressant treatment should be on stable doses for at least 6 months.
13. Patients who are taking systemic corticosteroids should be on a stable dose for at least 4 weeks.
14. Patients on anticoagulant therapy should be well-controlled prior to entry.
15. Patients taking iron and/or folic acid supplements should be on a stable dose for at least 4 weeks

Exclusion Criteria:

1. Patients whose mean haemoglobin level over the previous 12 months prior to screening was greater than 105 g/L (10.5g/dL)
2. Severe bone marrow failure
3. Patients with a platelet count of ≤ 70 x 109/L
4. Patients with known or suspected acquired somatic mutations affecting the bone marrow (e.g. acute myeloid leukaemia) which may be associated with PNH
5. Chemotherapy within 3 months of screening visit
6. History of recurrent bacterial infections or suspicion of active bacterial infections requiring antibiotic therapy
7. Planned or actual pregnancy or breast feeding (females)
8. Known allergy to ticks or severe reaction to arthropod venom (e.g. bee or wasp venom)
9. Unresolved N. meningitidis infection.
10. Patients who are not willing to receive adequate immunisation against N. meningitidis unless, in the opinion of the investigator, the risks of delaying therapy outweigh the risks of developing a meningococcal infection
11. Impaired hepatic function unless, in the opinion of the investigator, the risks of delaying therapy outweigh the risks of treatment in the presence of impaired hepatic function
12. Patients with a glomerular filtration rate (GFR) of <30mL/min/1.73m2 unless, in the opinion of the investigator, the risks of delaying therapy outweigh the risks of treatment in the presence of impaired renal function
13. Participation in other clinical trials within 4 weeks of signing the consent form
14. History of active systemic autoimmune diseases.
15. Any other systemic disorders that could interfere with the evaluation of the study treatment
16. Failure to comply with protocol requirements
17. Known Hepatitis B or Hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
HB (Haemoglobin) stabilisation rate and the avoidance of packed red blood cells (PRBC) transfusions | 9 months
  Haemoglobin stabilisation rate defined as haemoglobin greater than the set point for each patient during the pre-study randomisation period and the avoidance of PRBC transfusions during the treatment period.

SECONDARY OUTCOMES:
Number of units of packed red blood cells (PRBC) transfused | Day 1 to Day 180
  Number of units of packed red blood cells (PRBC) transfused from Baseline Day 1 to Day 180
Percentage of patients who achieve transfusion avoidance | Day 1 to Day 180
  Percentage of patients who achieve transfusion avoidance
Change in (QOl) Quality of Life score | Day 1 to Day 180
  Change in Quality of Life score
AUC (LDH) | Day 1 to Day 180
  AUC (Area under the curve) (LDH) Lactate Dehydrogenase
CH50 | Day 1 to Day 180
  CH50 (Classical haemolytic 50% lysis)

CONTACTS AND LOCATIONS:
Overall Officials: Andrius Degulys, MBBS, Principal Investigator — Vilnius University Hospital Santaros Klinikos
Locations (3):
- Almaty City Hospital No.7, Almaty, Microdistrict Kalkaman, Kazakhstan
- Vilnius University Hospital Santaros Klinikos , Santariškių St. 2, LT-08661,, Vilnius, Lithuania
- University of Kelaniya, Faculty of Medicine, Thalagolla Road, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: No